CLINICAL TRIAL: NCT07111832
Title: A Phase III, Multicenter, Randomized, Open-label, Active-controlled Study of SHR-A1811 Plus SHR-1316 Versus Toripalimab Plus Nab-paclitaxel in PD-L1-positive Locally Recurrent Unresectable or Metastatic Triple-negative Breast Cancer
Brief Title: A Clinical Trial of SHR-A1811 in the Treatment of Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-313
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: PD-L1-positive Locally Recurrent Unresectable or Metastatic Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Injections; toripalimab; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 and SHR-1316 Group (Experimental)
  Interventions: Drug: SHR-A1811 for Injection; Drug: SHR-1316 Injection
- Toripalimab and Nab-paclitaxel Group (Active Comparator)
  Interventions: Drug: Toripalimab Injection; Drug: Paclitaxel for Injection

INTERVENTIONS:
Drug: SHR-A1811 for Injection — SHR-A1811 for injection.
  Arms: SHR-A1811 and SHR-1316 Group
Drug: SHR-1316 Injection — SHR-1316 injection.
  Arms: SHR-A1811 and SHR-1316 Group
Drug: Toripalimab Injection — Toripalimab injection.
  Arms: Toripalimab and Nab-paclitaxel Group
Drug: Paclitaxel for Injection — Paclitaxel for injection.
  Arms: Toripalimab and Nab-paclitaxel Group

SUMMARY:
This study is to evaluate the progression-free survival (PFS) of SHR-A1811 combined with SHR-1316 in the first-line treatment of PD-L1-positive locally recurrent unresectable or metastatic triple-negative breast cancer with Toripalimab combined with Nab-paclitaxel, as assessed by blinded independent central review (BICR).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including both ends), female.
2. Pathologically confirmed locally recurrent unresectable or metastatic triple-negative breast cancer.
3. Expected survival ≥ 12 weeks.
4. Have adequate renal and hepatic function.
5. Patients voluntarily joined the study and signed the informed consent.

Exclusion Criteria:

1. Patients with active central nervous system (CNS) metastases who have not undergone surgery or radiotherapy.
2. Have other malignancies within the past 5 years.
3. Presence with uncontrollable third space effusion.
4. Have undergone other anti-tumor treatment within 4 weeks before the first dose.
5. A history of immunodeficiency.
6. Clinically significant cardiovascular diseases.
7. Known or suspected interstitial lung disease.
8. Known hereditary or acquired bleeding tendency.
9. Toxicities from prior anti-tumor therapy that have not recovered to ≤ Grade 1.
10. Known hypersensitivity to any of the study drugs or their excipients, or a history of allergy to humanized monoclonal antibody products.
11. Presence of other severe physical or mental disorders or clinically significant laboratory abnormalities.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | An average of 3 year.

SECONDARY OUTCOMES:
Overall response (OS) rate evaluated by investigators | An average of 3 year.
Clinical benefit rate (CBR) evaluated by investigators | An average of 3 year.
Duration of response (DoR) evaluated by investigators | An average of 3 year.
Progression-free survival on next-line therapy (PFS2) evaluated by investigators | An average of 3 year.
Adverse events (AEs) | An average of 3 year.
Serious adverse events (SAEs) | An average of 3 year.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital，Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided